CLINICAL TRIAL: NCT05163587
Title: Development of Low GI Composite Flour and Its Efficacy in Improving the Glycemic Profile in Type 2 Diabetes Patients _ A Randomized Clinical Trial.
Brief Title: Composite Flour and Its Antdiabetic Potential
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Sanaullah Iqbal, Chairman, Department of Food Science and Human Nutrition, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Composite flour
Record Dates: First submitted 2021-06-24; First posted 2021-12-20 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Blood Glucose, High; Body Weight Changes; Hyperlipidemias; Body Composition
Keywords: hyperglycemia; hyperlipidemia; weight control; diabetes type 2
MeSH Terms: conditions — Body Weight Changes; Hyperlipidemias; Hyperglycemia; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: two arm parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): control group will be provided with the commercially available whole-wheat flour for their consumption during the study period.
  Interventions: Combination Product: low GI composite flour
- Intervention (Experimental): intervention group will be provided with low GI composite flour for their chapatis during study period and they will be instructed to consume at least 4 chapatis each day.
  Interventions: Combination Product: low GI composite flour

INTERVENTIONS:
Combination Product: low GI composite flour — low GI composite flour orally in chapati form (3times/day)

SUMMARY:
A low glycemic multigrain flour for chapattis will be made from grains and cereals that are easily available in Pakistan. The nutritional profile and composition of test flour will be checked through proximate analysis method determined by AOAC. GI of test flour will be determined by comparing it with a reference food. The participants will be fed reference food i.e., 50gm glucose dissolved in 250ml water and test food serving having 50gm of available carbohydrates separately after an overnight fast. Finger prick method will be used to determine blood glucose levels at 0,15, 30, 45, 90 minutes. Trapezoidal rule will be used to determine iAUC and GI and GL will be determined by using standard formulas. Efficacy of test flour will be checked by human clinical trial. Control group will be fed chapatis made from test flour for 90 days. Anthropometry, body composition and biochemical measures including HbA1c, blood glucose (fasting and random) and lipid profile will be analyzed pre- and post-intervention and differences in their readings will be compared.

DETAILED DESCRIPTION:
The study comprises of four different phases.

* Phase 1: To develop a low GI composite flour.
* Phase 2: To assess nutritional profile and composition of the composite flour.
* Phase 3: To determine GI of chapatis made from test flour.
* Phase 4: Test the efficacy of test flour in improving glycemic profile through clinical trial.

Subjects: A total of 30 Type 2 diabetic patients aged between 30-60 years that are on oral medication will be selected for participation. They can be of either sex with no other complications of the disease. A written consent from the participants will be taken prior to study. Those participants who have insulin dependency, thyroid issues, are smokers and pregnant and lactating mothers will be excluded from the study. Prior to study, anthropometric measurements that will include height, weight, BMI, hip to waist ratio of each participant will be done. All the participants will complete testing for their HbA1c, lipid profile, fasting and random blood glucose measurements prior to study. For this, they will be called to University of Veterinary and Animal Sciences, Lahore for their blood sample collection. All the participants will be divided into two groups: control and intervention group with 15 participants in each group. The study will be conducted for 90 days and only those participants will be recruited that will be willing to complete the study duration with all the protocols for it. These include no major change in dietary pattern during the study. No change in physical activity i.e. doing any intense exercise or following any new workout routines. No change in medications or supplements during the study period is recommended.

Experimental design: The participants in the intervention group will be provided test flour for their chapattis (2kg for 10 days). The flour will be provided after each 10 days and they will be asked to use this flour for their chapattis. They will be guided to consume at least 3-4 chapattis each day while the participants in the control group will be asked to continue the flour, they are already using for their chapatti making. However during the study period all the participants will continue to follow their regular dietary habits, physical activity patterns and will continue taking their diabetes medication as per their schedule.

Biochemical testing: Along with the anthropometry, the participants will be tested biochemically by taking their blood samples at the start and at the end of the study. Before starting the trial, each participant will be tested for HbA1c and lipid profile. HbA1c tests will be done by Ion Exchange Resin method by using Glycohemoglobin HbA1 kit of brand Human Diagnostics. Lipid profile will also be checked at the baseline and after 3 months. For this purpose, Human diagnostic Kit will be used i.e. cholesterol liquicolor kit for cholesterol assessment, HDL cholesterol kit by Human diagnostics for HDL measurement, LDL liquicolor kit and TG Liquicolor mono kit by Human Diagnostics for LDL and triglycerides assessment. Random and Fasting blood glucose levels will be checked after every 10 days by using finger prick method through Glucometer (ACCU-CHECK® Performa Nano, Mannhim, Germany). For their interpretation, Guidelines of National Cholesterol Education Program (NCEP), (2004) will be used.

Statistical analysis: Statistical Package for Social Science software ( version 22) will be used for data analysis. Independent t test will be applied to check the differences between control and intervention groups. Paired t test will be used to determine differences among groups at initial and final time points within a group and their association will be checked at significance level of <0.05. Repeated measure design will be used to compare the blood glucose levels after every 10 days.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients of either sex that are non insulin dependent between age 30-60 years that are on oral medication only

Exclusion Criteria:

* patients with biochemical evidence of other diseases, thyroid patients, pregnant and lactating mothers and those above the age of 60 years or those who use insulin to control their blood glucose levels

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
hbA1c | 90 days
  by using low GI composite flour, the blood glucose levels of patients with type 2 diabetes should be controlled in a better way that can be determined by their hbA1c test value in 90 days
blood glucose levels | weekly
  by incorporating low GI food in daily meals will help lower the readings of daily blood glucose levels in patients with type 2 diabetes
lipid profile | 90 days
  lipid profile of patients with type 2 diabetes will be improved

SECONDARY OUTCOMES:
body weight | 90 days
  by keeping blood glucose levels in control and incorporating high fiber multigrain flour, it is expected that body weight of diabetic type 2 patients will be controlled in better way.
body composition | 90days
  body composition of participants will be measured through BIA

CONTACTS AND LOCATIONS:
Overall Officials: Azka Adeeb Alvi, Mphil, Principal Investigator — University of Veterinary and Animal Sciences
Locations (1):
- University of Veterinary and Animal Sciences, Paksitan, Lahore, Punjab Province, Pakistan